CLINICAL TRIAL: NCT01093911
Title: A Randomized, Double-blind, Placebo-controlled, Single-dose, Dose-escalating Study to Evaluate Safety, Tolerability, Pharmacokinetics, Immunogenicity and to Explore the Pharmacodynamics of CDP7657 Administered in Healthy Subjects and in SLE Patients.
Brief Title: Safety Study of CDP7657 in Healthy Volunteers and Patients With Systemic Lupus Erythematosus (SLE)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: SL0013; 2009-013617-10 (EudraCT Number)
Record Dates: First submitted 2010-03-12; First posted 2010-03-26 (Estimated); Last update posted 2013-01-04 (Estimated); Status verified 2013-01

CONDITIONS: Immune System Diseases; Autoimmune Diseases; Lupus Erythematosus, Systemic; Skin and Connective Tissue Diseases; Connective Tissue Disease
Keywords: Lupus; SLE
MeSH Terms: conditions — Immune System Diseases; Autoimmune Diseases; Lupus Erythematosus, Systemic; Skin and Connective Tissue Diseases; Connective Tissue Diseases | interventions — dapirolizumab pegol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- CDP7657 (Experimental): CDP7657 in dose escalating cohorts
  Interventions: Biological: CDP7657
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: CDP7657 — Ascending single doses of CDP7657
  Arms: CDP7657
Other: Placebo — Placebo: 0.9% sodium chloride aqueous solution
  Arms: Placebo

SUMMARY:
To evaluate safety, tolerability, pharmacokinetics and immunogenicity of CDP7657

ELIGIBILITY:
Inclusion Criteria:

* Healthy Volunteers and subjects with SLE

Exclusion Criteria:

* Severe neuropsychiatric or severe renal SLE
* History of chronic, recurrent, or recent severe infection
* Significant hematologic abnormalities
* History of cancer, heart failure, renal disease, liver disease or other serious illness

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2010-03; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Assessment of safety of CDP7657 as per Adverse Event (AE) reporting | Day 0 to 119

SECONDARY OUTCOMES:
Maximum plasma concentration (Cmax) | Day 0 to 119
Time corresponding to Cmax (Tmax) | Day 0 to 119
Terminal elimination half-life (t 1/2) | Day 0 to 119
Plasma levels of anti-CDP7657 antibodies | Day 0 to 119

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)
Locations (8):
- 6, Leuven, Belgium
- 9, Sofia, Bulgaria
- Germany (6):
  - 1, Berlin
  - 2, Erlangen
  - 3, Frankfurt
  - 4, Hanover
  - 8, Kiel
  - 7, Münster

REFERENCES:
- [Derived] Tocoian A, Buchan P, Kirby H, Soranson J, Zamacona M, Walley R, Mitchell N, Esfandiari E, Wagner F, Oliver R. First-in-human trial of the safety, pharmacokinetics and immunogenicity of a PEGylated anti-CD40L antibody fragment (CDP7657) in healthy individuals and patients with systemic lupus erythematosus. Lupus. 2015 Sep;24(10):1045-56. doi: 10.1177/0961203315574558. Epub 2015 Mar 16. PMID 25784719